CLINICAL TRIAL: NCT04585893
Title: LCCC 1950 - Rituximab for Multicentric Castleman Disease in Malawi, A Single-Arm Phase II Safety/Efficacy Trial
Brief Title: Safety and Efficacy of Rituximab for Treatment of Multicentric Castleman Disease in Malawi
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 1950; K01TW011470 (NIH)
Record Dates: First submitted 2020-09-10; First posted 2020-10-14 (Actual); Results first posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Multicentric Castleman Disease
Keywords: Multicentric Castleman Disease; MCD; HIV; Rituximab; single arm phase 2; safety and efficacy
MeSH Terms: conditions — Multi-centric Castleman's Disease; Macular dystrophy, corneal type 1 | interventions — Rituximab; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm Rituximab (Experimental): The safety and efficacy of first-line rituximab will be assessed through a risk-stratified rituximab-based Multicentric Castleman disease (MCD) The planned sample size is 27 adult patients accrued at a rate of 10 patients annually.
  High-risk patients (defined as patients with ECOG performance status >2 or hemoglobin <8 g/dL) will receive four weekly doses of rituximab (375 mg/m2) and etoposide (100 mg/m2).
  Low-risk patients will receive the same dose of rituximab (four weekly doses at 375 mg/m2) alone.
  Interventions: Drug: Rituximab; Drug: Etoposide

INTERVENTIONS:
Drug: Rituximab — 375 mg/m^2 administered via IV infusion weekly for four weeks. Administered via slow IV infusion, starting at 50mg/hr and increasing by 50mg/hr every 30 minutes to a maximum infusion rate of 400mg/hr.
  Other Names: Rituxan
Drug: Etoposide — Subjects with high-risk disease will receive 100 mg/m^2 etoposide weekly for four weeks administered over one hour via IV infusion after completion of rituximab
  Other Names: Toposar; VP-16

SUMMARY:
The purpose of this study is to determine the safety and efficacy of first-line, risk-stratified Rituximab-based Multicentric Castleman Disease (MCD) treatment in Malawi in a single-arm, phase II clinical trial. This study also aims to compare the cost-effectiveness of first-line Rituximab treatment for MCD in Malawi to chemotherapy.

DETAILED DESCRIPTION:
This study aims to determine the safety and efficacy of first-line, risk-stratified rituximab-based MCD treatment in Malawi in a single-arm, phase II clinical trial. The investigators will enroll 27 subjects with newly diagnosed or previously treated MCD (who have not previously received rituximab) requiring treatment (B symptoms or hemoglobin <10 g/dL). Subjects will be treated with four weekly doses of rituximab. High-risk subjects (defined as patients with Eastern Cooperative Oncology Group (ECOG) performance status >2 or hemoglobin <8 g/dL) will also receive etoposide chemotherapy. Subjects will be followed for one year for toxicity and two years for survival. The primary outcome will be safety, defined as the frequency of ≥Grade 3 treatment-related Common Terminology Criteria for Adverse Events (AEs). Secondary outcomes will be event-free survival (death, progression, or development of NHL) and 1- and 2-year overall survival (OS). The investigators also aim to compare the cost-effectiveness of first-line rituximab treatment for MCD in Malawi to chemotherapy (using the investigators' historical controls).

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed or previously treated subjects with KSHV-associated MCD that is pathologically confirmed by characteristic histologic features and latency-associated nuclear antigen (LANA) positivity by Immunohistochemistry (IHC).
2. Age is greater than or equal 18 years old at time of consent.
3. Can provide informed consent.
4. HIV-infected or HIV-uninfected.
5. If HIV-infected, must be on or willing to start antiretroviral therapy including lamivudine or tenofovir.
6. Willing to comply with study visits.
7. MCD treatment indicated based on the presence of a symptomatic MCD flare, defined as the presence of each of the following three criteria:

   1. Fever (subjective or objective)
   2. Lymphadenopathy or hepatosplenomegaly
   3. At least one of the following signs or symptoms attributable to MCD by the local study investigator:

      * Weight loss >5%
      * Malaise
      * Anemia (Hemoglobin <10 g/dL) within the past 4 weeks
      * Thrombocytopenia (Platelets <100 x 103/mL) NOTE: If only two of the three criteria are present, but the provider feels treatment is indicated for a symptomatic MCD flare, this will be allowed after communication with the study principal investigator (PI).

   Subjects with low hemoglobin within the past 4 weeks that have since received a blood transfusion are still eligible for participation. The subject's pre-transfusion hemoglobin value will be considered when determining risk classification.
8. Females of childbearing potential must have a negative urine pregnancy test within three days prior to registration.

   NOTE: Females are considered of childbearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months. Documentation of postmenopausal status must be provided.
9. Females must agree to abstain from breastfeeding during therapy and for 6 months after the completion of therapy.
10. Females of childbearing potential must be willing to abstain from heterosexual activity or to use two forms of effective methods of contraception from the time of informed consent until 12 months after treatment discontinuation. The two contraception methods can be comprised of two barrier methods, a barrier method plus a hormonal method, or an intrauterine device that meets <1% failure rate for protection from pregnancy in the product label.
11. Male subjects with female partners must have had a prior vasectomy or agree to use an adequate method of contraception (i.e., double barrier method: condom plus spermicidal agent) starting with the first dose of study therapy through 6 months after the last dose of study therapy.
12. More than 7 days without corticosteroid use prior to starting the treatment.

Exclusion Criteria:

1. Symptomatic, extensive-stage KS (T1 by the AIDS Clinical Trials Group (ACTG) staging system; T1 includes ulceration or edema from KS, raised or non-hard palate oral lesions, or any visceral involvement) requiring urgent treatment, to avoid potential rituximab-induced KS worsening.
2. Previous rituximab use for MCD.
3. Second active malignancy requiring systemic therapy.
4. If HIV negative and a) hepatitis B virus surface antigen positive or b) a combination of HepB core antibody positive and HepB surface antibody negative (indicative of chronic infection) unless on tenofovir or lamivudine. All HIV-infected patients must be on tenofovir or lamivudine as part of the inclusion criteria.
5. Active infection requiring systemic therapy.
6. Treatment with any investigational drug within 28 days prior to registration.
7. More than 7 days of corticosteroids immediately prior to enrollment. If the subject is taking corticosteroids for more than 7 days, they require a 7 day washout period before enrollment.
8. Bilirubin >3 mg/dL.
9. Creatinine clearance <30 ml/min by Cockcroft-Gault formula.
10. ECOG performance status >3.
11. Pregnant or breastfeeding (Note: Breast milk cannot be stored for future use while the mother is being treated in the study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2026-06-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Painschab, MD, Principal Investigator — University of North Carolina
Locations (1):
- UNC Project, Kamuzu Central Hospital, Lilongwe, Malawi

REFERENCES:
- See also: UNC Lineberger Comprehensive Cancer Center Website Homepage — https://unclineberger.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 06/22/2021 through 06/07/2024 at one center in Malawi.
Pre-assignment Details: Fifteen subjects were enrolled in the study between 06/22/2021 and 06/07/2024.
Groups:
- High-risk Patients: High-risk patients (defined as patients with ECOG performance status >2 or hemoglobin <8 g/dL) will receive four weekly doses of rituximab (375 mg/m2) and etoposide (100 mg/m2)..
- Low-risk Patients: Low-risk patients will receive the same dose of rituximab (four weekly doses at 375 mg/m2) alone.
Period: Overall Study
Arm/Group | High-risk Patients | Low-risk Patients
Started | 9 | 6
Completed | 8 | 6
Not Completed | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High-risk Patients | Low-risk Patients | Total
Number analyzed (Participants) | 9 | 6 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.44 (11.13) | 38.66 (8.23) | 39.73 (9.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 6 | 4 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 6 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 6 | 15
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Malawi | 9 | 6 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participant With Non-hematologic Grade ≥3 Adverse Events (AEs)
Description: Safety was assessed by the number of participants with non-hematologic Grade ≥3 adverse events (AEs) and treatment-related mortality. AEs were evaluated using the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE v5). CTCAE defines AE severity as: Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe or medically significant), Grade 4 (life-threatening), and Grade 5 (death related to AE).
Time Frame: From the start of rituximab-based therapy to 12 weeks. (Up to 13 weeks)
Population: All participants started the study.
Measure: Count of Participants; unit: Participants
Arm/Group | High-risk Patients | Low-risk Patients
Number analyzed (Participants) | 9 | 6
Participants | 0 | 0

2. Secondary Outcome: Characterization of MCD Presentation in Malawi
Description: Characterization of Multicentric Castleman disease (MCD) presentation in Malawi will be summarized using baseline demographics and laboratory values. Descriptive statistics will be performed.
Time Frame: Baseline - until 21 days
Reporting Status: Not Posted

3. Secondary Outcome: Overall Survival
Description: Overall survival is the measure of time from the first treatment day to the date of death for any cause. Subjects who have not had an event will be censored at the date of the last assessment documenting the subject was alive.
Time Frame: 90 days, 1 year, and 2 years
Reporting Status: Not Posted

4. Secondary Outcome: Event-free Survival
Description: Event-free survival is the measure of time after treatment during which no sign of cancer (refractory disease, relapse, non-Hodgkin lymphoma development, or death ) is found.
Time Frame: 90 days, 1 year, and 2 years
Reporting Status: Not Posted

5. Secondary Outcome: Efficacy of Risk-adjusted Treatment
Description: The efficacy of risk-adjusted treatment will be defined as the clinical response rate which is the resolution of presenting signs/symptoms that defined the Multicentric Castleman disease (MCD) attack. MCD attack/flare is defined as the presence of each of the following three criteria: 1) Fever (subjective or objective), 2) Lymphadenopathy or hepatosplenomegaly, 3) At least one of the following signs or symptoms attributable to MCD by the local study investigator: a) Weight loss >5%, b) Malaise, c) Anemia (Hemoglobin <10 g/dL), and d) Thrombocytopenia (Platelets <100 x 10^3/uL).
Time Frame: At the end of the treatment, 12 weeks after start of the treatment
Reporting Status: Not Posted

6. Secondary Outcome: Clinical Response Rate
Description: Clinical Response Rate will be defined as the percentage of subjects who achieved resolution of presenting signs/symptoms that defined the Multicentric Castleman disease (MCD) attack) without relapse.
Time Frame: At the end of the treatment, 12 weeks after start of the treatment
Reporting Status: Not Posted

7. Secondary Outcome: Radiological Response Rate
Description: The Radiological Response Rate will be defined as the percentage of subjects without relapse defined using chest radiography, abdominal sonography, and physical exam for gross lymphadenopathy.
  Response criteria for lymph node response will be Complete response (CR)- the disappearance of all evident disease; Partial response (PR)-at least a 50% decrease in target lesions with no increase in non-target lesions, Stable disease (SD)- Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD); PD- the appearance of a new lesion or at least a 50% increase in lesion size.
Time Frame: At the end of the treatment, 12 weeks after start of the treatment
Reporting Status: Not Posted

8. Secondary Outcome: Additional Safety
Description: Additional Safety will be defined as all Adverse Events occurred. AEs will be evaluated using National Cancer Institute's Common Terminology Criteria for Adverse Events version 5 (CTCAE v5).
Time Frame: First day of the treatment through 12 weeks (Up to 13 weeks)
Reporting Status: Not Posted

9. Secondary Outcome: The Rate of Kaposi Sarcoma Exacerbation
Description: The rate of Kaposi sarcoma exacerbation will be determined by symptomatic or clinical (dermatologic or visceral organ) exacerbation of the disease. All disease flares will be biopsy confirmed whenever possible.
Time Frame: Up to 2 years
Reporting Status: Not Posted

10. Secondary Outcome: Quality of Life- Patient-reported Outcomes Questionnaires
Description: Quality of Life- patient-reported outcomes (PRO) questionnaires will be assessed by the Patient-Reported Outcomes Measurement Information System Global Health Survey (PROMIS Global-10). The survey includes 10 items about mental and physical health rated on Likert scales ranging from 1 to 5, with higher scores indicative of better health.
Time Frame: Baseline, week3, end of the treatment, 12 weeks, 6 months after the treatment, 24 months after the treatment, time of relapse.
Reporting Status: Not Posted

11. Secondary Outcome: Change in Hemoglobin Measurement
Description: Hemoglobin will be measured in grams per deciliter (g/dL) at baseline, day 15, and end-of-treatment. Differences will be compared by paired t-test.
Time Frame: Baseline, Day 15 and End of treatment (approximately 6 weeks)
Reporting Status: Not Posted

12. Secondary Outcome: Change in Platelet Count Measurement
Description: Platelet count will be measured in microliters (µl) at baseline, day 15, and end-of-treatment. Differences will be compared by paired t-test.
Time Frame: Baseline, Day 15 and End of treatment (approximately 6 weeks)
Reporting Status: Not Posted

13. Secondary Outcome: Change in C-reactive Protein Measurement
Description: C-reactive protein (CRP) will be measured in milligrams per milliliter (mg/mL) at baseline, day 15, and end-of-treatment. Differences will be compared by paired t-test.
Time Frame: Baseline, Day 15 and End of treatment (approximately 6 weeks)
Reporting Status: Not Posted

14. Secondary Outcome: Change in Kaposi Sarcoma Herpesvirus Viral Load Measurement
Description: Kaposi sarcoma herpesvirus (KSHV) viral load will be measured in copies per milliliter (copies/mL) at baseline, day 15, and end-of-treatment. Differences will be compared by paired t-test.
Time Frame: Baseline, Day 15 and End of treatment (approximately 6 weeks)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 12 weeks
Description: Adverse events were collected from day one of the study drug administration to 30 days after completion of treatment.
Arm/Group | High-risk Patients | Low-risk Patients
All-Cause Mortality (participants affected / at risk) | 1/9 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/9 | 1/6
Other Adverse Events (participants affected / at risk) | 9/9 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High-risk Patients (N=9) | Low-risk Patients (N=6)
Anemia (Blood and lymphatic system disorders) | 1 | 0
neutrophil count decreased (Blood and lymphatic system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High-risk Patients (N=9) | Low-risk Patients (N=6)
Anemia (Blood and lymphatic system disorders) | 8 | 5
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Flu like symptoms (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 2 | 0
Lung infection (Infections and infestations) | 4 | 0
Blood bilirubin increased (Investigations) | 1 | 1
Blood lactate dehydrogenase increased (Investigations) | 4 | 0
Creatinine increased (Investigations) | 3 | 1
Lymphocyte count decreased (Investigations) | 7 | 1
Neutrophil count decreased (Investigations) | 5 | 1
Hypoalbuminemia (Investigations) | 3 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypotension (Vascular disorders) | 2 | 0
Alkaline Phosphatase Increased (Investigations) | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 0 | 1
Bruising (Injury, poisoning and procedural complications) | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0
Fever (General disorders) | 2 | 1
Hypertension (Vascular disorders) | 1 | 0
Laryngeal Inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Platelet count decreased (Blood and lymphatic system disorders) | 2 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-20): https://cdn.clinicaltrials.gov/large-docs/93/NCT04585893/Prot_SAP_000.pdf